CLINICAL TRIAL: NCT01529528
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled, Therapeutic Confirmatory Trial(Phase 3) to Evaluate Efficacy and Safety of CWP-0403 in Type 2 DM Patients
Brief Title: A Study to Efficacy and Safety of CWP-0403 in Type 2 Diabetes Mellitus Patients
Acronym: CWP-DIANA-301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CWP-DIANA-301
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: CWP-0403; type 2 DM; Efficacy; Safety; Phase 3
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — anagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo of CWP-0403 100mg (Placebo Comparator): Placebo of CWP-0403 100mg
  Interventions: Drug: Placebo of Anagliptin
- CWP-0403 200mg (Experimental): CWP-0403 200mg
  Interventions: Drug: Anagliptin
- CWP-0403 100mg (Experimental): CWP-0403 100mg
  Interventions: Drug: Anagliptin

INTERVENTIONS:
Drug: Anagliptin — Anagliptin 100mg, tablet, BID
  Arms: CWP-0403 100mg
Drug: Anagliptin — Anagliptin 100mg, tablet, BID
  Arms: CWP-0403 200mg
Drug: Placebo of Anagliptin — Placebo of Anagliptin 100mg, tablet, BID
  Arms: Placebo of CWP-0403 100mg

SUMMARY:
This trial is to evaluate the efficacy and safety of CWP-0403 at 100 mg or 200 mg twice daily compared with placebo in type 2 diabetic patients with inadequate glycemic control by diet therapy or combination of diet and exercise therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM patients
* Subjects who couldn't control the blood glucose despite of a dietary and exercise therapy more than 6 weeks at screening visit
* FPG ≤ 270mg/dL at screening visit
* Patients who consent to participate in this trial by written Informed Consent Form

Exclusion Criteria:

* Type 1 DM or secondary diabetes
* Subjects who are administrating insulin or need to insulin therapy
* History of oral anti-hyperglycemic drugs within 6 weeks before screening visit
* Body mass index < 20 kg/m2 or > 40.0kg/m2
* Subjects who are assessed to be inappropriate for this trial by investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The Change in HbA1c from baseline to week24 | 0wk, 8wk, 16wk, 24wk

SECONDARY OUTCOMES:
The proportion of subjects achieving HbA1c<6.5% at week24 | 0wk, 8wk, 16wk, 24wk
The proportion of subjects achieving HbA1c<7% at week24 | 0wk, 8wk, 16wk, 24wk
The change from baseline to week 24: Fasting plasma glucose | 0wk, 24wk
change from baseline to week 24 in Fasting serum insulin | 0 wk, 24 wk
change from baseline to week 24 in Fasting serum pro-insulin | 0 wk, 24wk
change in from baseline to week 24 fasting serum c-peptide | 0wk, 24wk
change from baseline to week 24 in HOMA-β | owjm 24wk
change from baseline to week 24 in HOMA-IR | 0wk, 24 wk

CONTACTS AND LOCATIONS:
Overall Officials: Sung Woo Park, M.D., PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea